CLINICAL TRIAL: NCT05998902
Title: Trophic Enteral Feeding Combined With Supplemental Parenteral Nutrition Treatment in Patients With Severe Stroke (OPENS-2): a Multicentre, Prospective, Randomised, Open-label, Blinded-endpoint Trial
Brief Title: Optimizing Early Nutrition Support in Severe Stroke-2
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Wen Jiang-3 (Other)
Collaborators: Tang-Du Hospital (Other); Xi'an Central Hospital (Other); Xi'an Gaoxin Hospital (Other); First Affiliated Hospital Xi'an Jiaotong University (Other); Xi'an No.3 Hospital (Other Government); First People's Hospital of Xianyang (Other); Nanfang Hospital, Southern Medical University (Other); Tongji Hospital (Other); Qilu Hospital of Shandong University (Other); The Second Hospital of Shandong University (Other); PLA 960 Hospital (Unknown); Daping Hospital, The Third Military Medical University (Army Medical University) (Unknown); The Second Affiliated Hospital of Guangzhou University of Chinese Medicine (Unknown); First Hospital Affiliated to Zhengzhou University (Unknown); Gansu Provincial Central Hospital (Unknown); The First Hospital of Changsha City (Unknown); Shaanxi Provincial People's Hospital (Other); Yulin No.2 Hospital (Other); Yulin No.1 Hospital (Unknown); Xijing Hospital (Other)
Responsible Party: Sponsor-Investigator, Wen Jiang-3, Head of Neurology, Xijing Hospital
Organization: Xijing Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: XJLL-KY-20222214
Record Dates: First submitted 2023-07-26; First posted 2023-08-21 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Severe Stroke; Acute Stroke; Dysphagia
Keywords: Severe Stroke; Acute Stroke; Dysphagia; supplemental parenteral nutrition; trophic feeding; pneumonia
MeSH Terms: conditions — Stroke; Deglutition Disorders; Pneumonia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Full enteral feeding (Active Comparator): Patients will receive full enteral feeding through nasogastric tube or nasointestinal tube.
  Interventions: Procedure: Full enteral feeding
- Trophic enteral feeding combined with supplemental parenteral nutrition (Experimental): Patients will receive trophic enteral feeding combined with supplemental parenteral feeding.
  Interventions: Procedure: Trophic enteral feeding combined with supplemental parenteral nutrition

INTERVENTIONS:
Procedure: Trophic enteral feeding combined with supplemental parenteral nutrition — The caloric goal of the first day is one-third of caloric requirements, the second day is half of caloric requirements, the third day is 70-100% and sustained for 1 week. Patients will receive the trophic enteral feeding with a caloric target of 500kcal/d (20-35ml/h), and the remaining calories are supplemented by parenteral nutrition. Protein requirements are calculated at 1.2 to 1.5 g per kilogram of body weight per day.
  Arms: Trophic enteral feeding combined with supplemental parenteral nutrition
Procedure: Full enteral feeding — The caloric goal of the first day is one-third of caloric requirements, the second day is half of caloric requirements, the third day is 70-100% and sustained for 1 week. Protein requirements are calculated at 1.2 to 1.5 g per kilogram of body weight per day. Enteral nutrition is given through nasogastric tube or nasointestinal tube.
  Arms: Full enteral feeding

SUMMARY:
Post stroke pneumonia (PSP) is one of the common early complications of stroke. Post-stroke infections, in general, are associated with less favorable neurologic outcomes. Aspiration is one of the most feared complications of enteral nutrition and can lead to the occurrence of pneumonia. Severe stroke patients are at high risk for aspiration due to some factors such as the reduced level of consciousness, inability to protect the airway and so on. The purpose of this study is to explore the ideal nutrition support strategy for patient with acute severe stroke to help reduce the incidence of PSP and improve the prognosis.

DETAILED DESCRIPTION:
As one of the most common complication of stroke, some studies showed that post-stroke pneumonia (PSP) in stroke patients requiring intensive care is associated with an increase of ICU length of stay and hospital mortality and poorer functional outcomes in survivors. The peak period of PSP is within the first week after stroke. Aspiration and poor nutritional status are important factors leading to pneumonia in stroke patients. Compared with full enteral nutrition (EN), initial trophic enteral feeding was associated with less gastrointestinal intolerance and could reduce the rate of regurgitation. However, trophic enteral feeding could not meet the daily caloric needs and hypocaloric enteral nutrition might be associated with increased mortality. This study is designed to explore whether initial trophic enteral nutrition combined with supplemental parenteral nutrition (SPN) can help reduce the incidence of PSP and improve the prognosis in severe patients with stroke.

This study will enroll 546 severe stroke patients who meet the inclusion criteria. Upon admission to the ICU, patients will be randomly assigned at a 1:1 ratio into groups of full enteral feeding (controlled) and trophic enteral feeding combined with supplemental parenteral feeding (experimented) for 7 days.

ELIGIBILITY:
Inclusion Criteria:

1. Age≥18 years
2. Definite diagnosis of acute stroke (GCS ≤12 or NIHSS≥11)
3. The randomized nutritional treatment could be initiated up to 72 hours after symptom onset.
4. Any cases of profiles #3 through 5 in Water Swallowing Test or with disorder of consciousness.
5. Plan to receive nutritional support treatment for at least 7 days.
6. Informed consent.

Exclusion Criteria:

1. Receiving parenteral nutrition support
2. Contraindications of enteral nutrition
3. Complicated with the disease which only have life expectancy < 7 days
4. Admission with infection signs
5. Dementia or severe disability (mRS>4) before stroke
6. Antibiotics were used within the previous 7 days
7. Subarachnoid hemorrhage, cerebral arteriovenous malformation
8. Presence of coexisting medical conditions that could interfere with outcome assessment and/or follow-up (a. advanced cancer; b. severe pulmonary dysfunction [forced expiratory volume in 1 second < 50% or/and moderate to severe acute lung injury (PaO2/FiO2)<200mmHg]; c. cardiac insufficiency (NYHA class > I; cardiac structural and/or functional abnormalities such as EF< 50%, abnormal cardiac chamber enlargement, moderate/severe ventricular hypertrophy, or moderate/severe valvular stenosis); d. Severe liver failure [Child-Pugh score≥7]; e. Severe renal failure [glomerular filtration rate ≤30mL/min or serum creatinine ≥4mg/dL]
9. Currently participating in other clinical trial
10. Pregnant woman
11. Patient who is considered highly likely not to adhere to the study treatment or follow-up protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 546 (Estimated)
Dates: Start 2023-12-20 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of post stroke pneumonia | up to 7 days

SECONDARY OUTCOMES:
The time from randomisation to the onset of the post stroke pneumonia | up to 7 days
Daily calorie delivery | up to 7 days
Daily protein delivery | up to 7 days
Insulin utilization | up to 7 days
  Insulin utilization during the first 7 days post-randomization
The incidence of gastrointestinal complications | up to 7 days
  Vomiting, diarrhea, gastric retention, gastrointestinal bleeding
The use of prokinetic agents | up to 7 days
  The usage rate of prokinetic agents
The occurrence of infections | 1 day of ICU discharge
  The rate and onset time of infections from randomisation to ICU discharge
The length of ICU stay | 1 day of ICU discharge
Mortality | 1 day of ICU discharge
  from randomisation to all cause death during ICU stay.
The All-cause mortality rate | 28 days after enrollment
  from randomisation to all cause death at 28 days
Cardiac failure | 1 day of ICU discharge
  The incidence of cardiac failure from randomisation to ICU discharge
Tracheotomy | 1 day of ICU discharge
  The incidence of tracheotomy from randomisation to ICU discharge
Mechanical ventilation | 1 day of ICU discharge
  The incidence of mechanical ventilation from randomisation to ICU discharge
Continuous renal replacement therapy | 1 day of ICU discharge
  The incidence of continuous renal replacement therapy from randomisation to ICU discharge
The use of vasoactive agents | 1 day of ICU discharge
  The usage rate of vasoactive agents from randomisation to ICU discharge
Deep venous thrombosis | 1 day of ICU discharge
  The incidence of deep venous thrombosis from randomisation to ICU discharge
The score of National Institute of Health stroke scale at ICU discharge | 1 day of ICU discharge
  National Institute of Health stroke scale, with scores ranging from 0 (normal function) to 42 (functional impairment) was used to evaluate the impairment caused by a stroke.
Glasgow Coma Scale at ICU discharge | 1 day of ICU discharge
  Glasgow Coma Scale,with scores ranging from 3 (no response) to 15 (normal response), was used to grade the conscious state.
modified Rankin scale at ICU discharge | 1 day of ICU discharge
  modified Rankin scale score, with score ranging from 0 (normal) to 6 (death), was used to evaluate the functional outcomes after stroke.
modified Rankin scale | 90 days after enrollment
  modified Rankin scale score, with score ranging from 0 (normal) to 6 (death), was used to evaluate the functional outcomes after stroke, including ordinal mRS, excellent outcome (mRS 0-1), and functional independence (mRS 0-2)

OTHER OUTCOMES:
Composite endpoint of all-cause mortality and post-stroke pneumonia | 90 days after randomization
  Hierarchical composite endpoint of all-cause mortality and post-stroke pneumonia within 90 days
Composite endpoint of all-cause mortality and post-stroke pneumonia | 7 days after randomization
  Hierarchical composite endpoint of all-cause mortality and post-stroke pneumonia within 7 days
Time from randomization to the first occurrence of either all-cause death or post-stroke pneumonia | 90 days after randomization
  Time from randomization to the first occurrence of either all-cause death or post-stroke pneumonia within 90 days

CONTACTS AND LOCATIONS:
Locations (30):
- China (30):
  - Chongqing University Three Gorges Hospital, Chongqing, Chongqing Municipality
  - Daping Hospital, The Third Military Medical University, Chongqing, Chongqing Municipality
  - Gansu Provincal Central Hospital, Lanzhou, Gansu
  - Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong
  - The Second Affiliated Hospital of Guangzhou University of Chinese Medicine, Guangzhou, Guangdong
  - The Affiliated Hospital of Guizhou Medical University, Guiyang, Guizhou
  - First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Tongji Hospital, Wuhan, Hubei
  - The First Hospital of Changsha City, Changsha, Hunan
  - The Second Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - General Hospital of Ningxia Medical University, Yinchuan, Ningxia
  - Shaanxi Second Provincal People's Hospital, Xi'an, Shaanxi
  - Tangdu Hospital, Xi'an, Shaanxi
  - The first affiliated hospital of Xi'an Jiaotong University, Xi'an, Shaanxi
  - Xi'an Central Hospital, Xi'an, Shaanxi
  - Department of Neurology, Xijing Hospital, Xi'an, Shaanxi
  - Shannxi Provincal People's Hospital, Xi'an, Shaanxi
  - The First Affiliated Hospital of Xi'an Medical University, Xi'an, Shaanxi
  - Xi'an Gaoxin Hospital, Xi'an, Shaanxi
  - Xi'an No.3 Hospital, Xi'an, Shaanxi
  - Xianyang Hospital, Yan'an University, Xianyang, Shaanxi
  - The First People's Hospital of Xianyang, Xianyang, Shaanxi
  - Yulin No.1 Hospital, Yulin, Shaanxi
  - Yulin No.2 Hospital, Yulin, Shaanxi
  - Qilu Hospital of Shangdong University, Jinan, Shandong
  - The PLA 960 Hospital, Jinan, Shandong
  - The Second Hospital of Shandong University, Jinan, Shandong
  - Liaocheng People's Hospital, Liaocheng, Shandong
  - People's Hospital of Xinjiang Uygur Autonomous Region, Ürümqi, Xinjiang
  - The Second Affiliated Hospital of Xinjiang Medical University, Ürümqi, Xinjiang

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Meisel A, Smith CJ. Prevention of stroke-associated pneumonia: where next? Lancet. 2015 Nov 7;386(10006):1802-4. doi: 10.1016/S0140-6736(15)00127-0. Epub 2015 Sep 3. No abstract available. PMID 26343837
- [Background] Wilson RD. Mortality and cost of pneumonia after stroke for different risk groups. J Stroke Cerebrovasc Dis. 2012 Jan;21(1):61-7. doi: 10.1016/j.jstrokecerebrovasdis.2010.05.002. Epub 2010 Jun 17. PMID 22225864
- [Background] Kishore AK, Vail A, Chamorro A, Garau J, Hopkins SJ, Di Napoli M, Kalra L, Langhorne P, Montaner J, Roffe C, Rudd AG, Tyrrell PJ, van de Beek D, Woodhead M, Meisel A, Smith CJ. How is pneumonia diagnosed in clinical stroke research? A systematic review and meta-analysis. Stroke. 2015 May;46(5):1202-9. doi: 10.1161/STROKEAHA.114.007843. Epub 2015 Apr 9. PMID 25858238
- [Background] Suda S, Aoki J, Shimoyama T, Suzuki K, Sakamoto Y, Katano T, Okubo S, Nito C, Nishiyama Y, Mishina M, Kimura K. Stroke-associated infection independently predicts 3-month poor functional outcome and mortality. J Neurol. 2018 Feb;265(2):370-375. doi: 10.1007/s00415-017-8714-6. Epub 2017 Dec 16. PMID 29249057
- [Background] Cohen DL, Roffe C, Beavan J, Blackett B, Fairfield CA, Hamdy S, Havard D, McFarlane M, McLauglin C, Randall M, Robson K, Scutt P, Smith C, Smithard D, Sprigg N, Warusevitane A, Watkins C, Woodhouse L, Bath PM. Post-stroke dysphagia: A review and design considerations for future trials. Int J Stroke. 2016 Jun;11(4):399-411. doi: 10.1177/1747493016639057. Epub 2016 Mar 22. PMID 27006423
- [Background] Westendorp WF, Nederkoorn PJ, Vermeij JD, Dijkgraaf MG, van de Beek D. Post-stroke infection: a systematic review and meta-analysis. BMC Neurol. 2011 Sep 20;11:110. doi: 10.1186/1471-2377-11-110. PMID 21933425
- [Background] Finlayson O, Kapral M, Hall R, Asllani E, Selchen D, Saposnik G; Canadian Stroke Network; Stroke Outcome Research Canada (SORCan) Working Group. Risk factors, inpatient care, and outcomes of pneumonia after ischemic stroke. Neurology. 2011 Oct 4;77(14):1338-45. doi: 10.1212/WNL.0b013e31823152b1. Epub 2011 Sep 21. PMID 21940613
- [Background] de Montmollin E, Ruckly S, Schwebel C, Philippart F, Adrie C, Mariotte E, Marcotte G, Cohen Y, Sztrymf B, da Silva D, Bruneel F, Gainnier M, Garrouste-Orgeas M, Sonneville R, Timsit JF; OUTCOMEREA Study Group. Pneumonia in acute ischemic stroke patients requiring invasive ventilation: Impact on short and long-term outcomes. J Infect. 2019 Sep;79(3):220-227. doi: 10.1016/j.jinf.2019.06.012. Epub 2019 Jun 22. PMID 31238051
- [Background] Suntrup-Krueger S, Kemmling A, Warnecke T, Hamacher C, Oelenberg S, Niederstadt T, Heindel W, Wiendl H, Dziewas R. The impact of lesion location on dysphagia incidence, pattern and complications in acute stroke. Part 2: Oropharyngeal residue, swallow and cough response, and pneumonia. Eur J Neurol. 2017 Jun;24(6):867-874. doi: 10.1111/ene.13307. Epub 2017 Apr 27. PMID 28449405
- [Background] Al-Khaled M. The multifactorial etiology of stroke-associated pneumonia. J Neurol Sci. 2019 May 15;400:30-31. doi: 10.1016/j.jns.2019.02.042. Epub 2019 Mar 12. No abstract available. PMID 30884370
- [Background] McClave SA, DeMeo MT, DeLegge MH, DiSario JA, Heyland DK, Maloney JP, Metheny NA, Moore FA, Scolapio JS, Spain DA, Zaloga GP. North American Summit on Aspiration in the Critically Ill Patient: consensus statement. JPEN J Parenter Enteral Nutr. 2002 Nov-Dec;26(6 Suppl):S80-5. doi: 10.1177/014860710202600613. PMID 12405628
- [Background] Jabbar A, Chang WK, Dryden GW, McClave SA. Gut immunology and the differential response to feeding and starvation. Nutr Clin Pract. 2003 Dec;18(6):461-82. doi: 10.1177/0115426503018006461. PMID 16215082
- [Background] Singer P, Blaser AR, Berger MM, Alhazzani W, Calder PC, Casaer MP, Hiesmayr M, Mayer K, Montejo JC, Pichard C, Preiser JC, van Zanten ARH, Oczkowski S, Szczeklik W, Bischoff SC. ESPEN guideline on clinical nutrition in the intensive care unit. Clin Nutr. 2019 Feb;38(1):48-79. doi: 10.1016/j.clnu.2018.08.037. Epub 2018 Sep 29. PMID 30348463
- [Background] Uozumi M, Sanui M, Komuro T, Iizuka Y, Kamio T, Koyama H, Mouri H, Masuyama T, Ono K, Lefor AK. Interruption of enteral nutrition in the intensive care unit: a single-center survey. J Intensive Care. 2017 Aug 4;5:52. doi: 10.1186/s40560-017-0245-9. eCollection 2017. PMID 28794882
- [Background] Harvey SE, Parrott F, Harrison DA, Bear DE, Segaran E, Beale R, Bellingan G, Leonard R, Mythen MG, Rowan KM; CALORIES Trial Investigators. Trial of the route of early nutritional support in critically ill adults. N Engl J Med. 2014 Oct 30;371(18):1673-84. doi: 10.1056/NEJMoa1409860. Epub 2014 Oct 1. PMID 25271389
- [Background] Altintas ND, Aydin K, Turkoglu MA, Abbasoglu O, Topeli A. Effect of enteral versus parenteral nutrition on outcome of medical patients requiring mechanical ventilation. Nutr Clin Pract. 2011 Jun;26(3):322-9. doi: 10.1177/0884533611405790. Epub 2011 Apr 29. PMID 21531737
- [Background] Reignier J, Boisrame-Helms J, Brisard L, Lascarrou JB, Ait Hssain A, Anguel N, Argaud L, Asehnoune K, Asfar P, Bellec F, Botoc V, Bretagnol A, Bui HN, Canet E, Da Silva D, Darmon M, Das V, Devaquet J, Djibre M, Ganster F, Garrouste-Orgeas M, Gaudry S, Gontier O, Guerin C, Guidet B, Guitton C, Herbrecht JE, Lacherade JC, Letocart P, Martino F, Maxime V, Mercier E, Mira JP, Nseir S, Piton G, Quenot JP, Richecoeur J, Rigaud JP, Robert R, Rolin N, Schwebel C, Sirodot M, Tinturier F, Thevenin D, Giraudeau B, Le Gouge A; NUTRIREA-2 Trial Investigators; Clinical Research in Intensive Care and Sepsis (CRICS) group. Enteral versus parenteral early nutrition in ventilated adults with shock: a randomised, controlled, multicentre, open-label, parallel-group study (NUTRIREA-2). Lancet. 2018 Jan 13;391(10116):133-143. doi: 10.1016/S0140-6736(17)32146-3. Epub 2017 Nov 8. PMID 29128300
- [Background] Compher C, Bingham AL, McCall M, Patel J, Rice TW, Braunschweig C, McKeever L. Guidelines for the provision of nutrition support therapy in the adult critically ill patient: The American Society for Parenteral and Enteral Nutrition. JPEN J Parenter Enteral Nutr. 2022 Jan;46(1):12-41. doi: 10.1002/jpen.2267. Epub 2022 Jan 3. PMID 34784064
- [Background] Heidegger CP, Berger MM, Graf S, Zingg W, Darmon P, Costanza MC, Thibault R, Pichard C. Optimisation of energy provision with supplemental parenteral nutrition in critically ill patients: a randomised controlled clinical trial. Lancet. 2013 Feb 2;381(9864):385-93. doi: 10.1016/S0140-6736(12)61351-8. Epub 2012 Dec 3. PMID 23218813
- [Background] Shi J, Wei L, Huang R, Liao L. Effect of combined parenteral and enteral nutrition versus enteral nutrition alone for critically ill patients: A systematic review and meta-analysis. Medicine (Baltimore). 2018 Oct;97(41):e11874. doi: 10.1097/MD.0000000000011874. PMID 30313021
- [Background] National Heart, Lung, and Blood Institute Acute Respiratory Distress Syndrome (ARDS) Clinical Trials Network; Rice TW, Wheeler AP, Thompson BT, Steingrub J, Hite RD, Moss M, Morris A, Dong N, Rock P. Initial trophic vs full enteral feeding in patients with acute lung injury: the EDEN randomized trial. JAMA. 2012 Feb 22;307(8):795-803. doi: 10.1001/jama.2012.137. Epub 2012 Feb 5. PMID 22307571
- [Background] Zhao J, Yuan F, Song C, Yin R, Chang M, Zhang W, Zhang B, Yu L, Jia Y, Ma Y, Song Y, Wang C, Song C, Wang X, Shang L, Yang F, Jiang W; OPENS Trial Investigators. Safety and efficacy of three enteral feeding strategies in patients with severe stroke in China (OPENS): a multicentre, prospective, randomised, open-label, blinded-endpoint trial. Lancet Neurol. 2022 Apr;21(4):319-328. doi: 10.1016/S1474-4422(22)00010-2. Epub 2022 Feb 24. PMID 35219379